CLINICAL TRIAL: NCT01983748
Title: A NON-COMMERCIAL, MULTICENTER, RANDOMIZED, TWO-ARMED, OPEN-LABEL PHASE III STUDY TO EVALUATE THE ADJUVANT VACCINATION WITH TUMOR RNA-LOADED AUTOLOGOUS DENDRITIC CELLS VERSUS OBSERVATION OF PATIENTS WITH RESECTED MONOSOMY 3 UVEAL MELANOMA
Brief Title: Dendritic Cells Plus Autologous Tumor RNA in Uveal Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Collaborators: University Hospital Lübeck (Other); University Hospital Munich (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Homburg/Saar (Unknown); Universitätsklinikum Köln (Other); University Hospital Tuebingen (Other); University Hospital, Essen (Other); Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, PD Dr. med. univ. Beatrice Schuler-Thurner, Coordinating Investigator, University Hospital Erlangen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DERMA-ER-DC 08
Record Dates: First submitted 2013-09-17; First posted 2013-11-14 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-03

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma, Monosomy 3
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Biological/Vaccine; Autologous Dendritic Cells loaded with autologous Tumor RNA
  Interventions: Biological: Autologous Dendritic Cells loaded with autologous Tumor RNA
- B (No Intervention): Control, Standard of care, which is clinical control every 3 months

INTERVENTIONS:
Biological: Autologous Dendritic Cells loaded with autologous Tumor RNA
  Arms: A

SUMMARY:
Patients suffering from uveal melanoma (typed positive for monosomy 3 and without evidence for metastases) will be vaccinated over a period of 2 years with Dendritic Cell loaded with autologous Tumor RNA.

200 patients will be included. The Trial is an open multicenter Phase III Trial.

DETAILED DESCRIPTION:
Trial arm A (DCaT-RNA) = Experimental intervention: Patients in arm A receive 8 vaccinations over a period of 2 years consisting of autologous, mature, monocyte-derived Dendritic Cells loaded with autologous tumor RNA (20 mio DC per vaccination); cells are given via intravenous infusions; vaccinations are followed by a 1 year observation (staging every 3 months)

Trial arm B (Observation) = Control: Patients in arm B receive standard care (observation only with staging every 3 months)

ELIGIBILITY:
Inclusion Criteria:

* Patients must suffer from melanoma of the uvea (stage T2, T3 and T4 [AJCC TNM grading 2009]).
* Uveal melanoma must be resected and display a monosomy for chromosome 3 (will be determined by a validated qualitative analysis of loss of heterozygosity). Tumor material has to be stored appropriately in RNAlater solution for RNA preparation.
* The patient has to be free of detectable tumor at the time point of study enrollment (adjuvant setting), as assessed by clinical inspection, abdominal sonography, chest X-ray and evaluation of the tumor-marker S-100..
* Patients must have a WHO performance status of 0, 1 or 2 and must be in stable medical condition.
* Patients must be between 18 and 75 years old and must be able and willing to give informed consent.
* Women of child-bearing age must have a negative pregnancy test, and must oblige to use effective contraception until at least 4 weeks after the last vaccination.
* Patients must be willing to get hospitalized for at least 4 hours following vaccination(s), and to cooperate for the whole period of the trial.
* Patients must have fully recovered from surgery.
* Signed informed consent

Exclusion Criteria:

* Any other major serious illness [e.g. active systemic infections, immunodeficiency disease, clinically significant heart disease, respiratory disease, bleeding disorders, cancer etc.] or a contraindication to leukapheresis.
* Evidence for HIV-1, HIV -2, HTLV-1, HBV, or HCV infection.
* Active autoimmune disease (such as but not limited to Lupus erythematosus, autoimmune thyroiditis or uveitis, multiple sclerosis, inflammatory bowel disease). Vitiligo and pathological laboratory results (autoantibodies) without clinical symptoms are, however, not an exclusion criterion.
* Previous splenectomy or radiation therapy to the spleen.
* Patients with organ allografts.
* Concomitant treatment with chemotherapy, immunotherapy, any investigational drug and paramedical substances. Patients may receive concomitant medications to control symptoms such as analgetics, antihypertensive medication, etc.
* History of other active malignant neoplasm within the preceding 5 years (excluding non-melanoma skin cancer or carcinoma in situ of the cervix).
* Organic brain syndrome or significant psychiatric abnormality which would impede informed consent and / or AND preclude participation in the full protocol and follow up.
* Positive pregnancy test / Pregnancy or lactation. If pregnancy occurs during the course of the trial to female patients in arm A or B, the patient has to be excluded.
* Detection of metastases. If uveal melanoma metastases appear during the course of the trial, the patient has to be excluded.
* Lack of compliance of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08-05 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Prolongation of Overall survival | Assessment every 3 months
  Clinical staging every 3 months from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months, followed by telephone interviews.

SECONDARY OUTCOMES:
Prolongation of disease free survival | Assessment every 3 months
  Skin, lymph node and ophtalmological inspection , medical history, laboratory, and abdominal sonography will be performed every 3 months, chest x ray will be performed every 6 months

OTHER OUTCOMES:
Assessment for induction of immune responses | The induction of immune responses will be researched in selected patients (in a minimum of 15 survivors per trial arm) 2 years after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Schuler-Thurner, MD, Principal Investigator — University Hospital Erlangen
Locations (8):
- Germany (8):
  - Dept. of Dermatology, University Hospital, Erlangen, Bavaria
  - University Hospital Department of Ophtalmology, Erlangen, Bavaria
  - University Hospital Department of Ophtalmology, Würzburg, Bavaria
  - Städtisches Klinikum, Dessau
  - University Hospital Department of Ophtalmology, Essen
  - University Hospital Department of Ophtalmology, Homburg/Saar
  - University Hospital Department of Ophtalmology, Lübeck
  - University Hospital Department of Ophtalmology, Tübingen

REFERENCES:
- [Background] Schuler-Thurner B, Bartz-Schmidt KU, Bornfeld N, Cursiefen C, Fuisting B, Grisanti S, Heindl LM, Holbach L, Keseru M, Knorr H, Koch K, Kruse F, Meiller R, Metz C, Meyer-ter-Vehn T, Much M, Reinsberg M, Schliep S, Seitz B, Schuler G, Susskind D, Viestenz A, Wagenfeld L, Zeschnigk M. [Immunotherapy of uveal melanoma: vaccination against cancer. Multicenter adjuvant phase 3 vaccination study using dendritic cells laden with tumor RNA for large newly diagnosed uveal melanoma]. Ophthalmologe. 2015 Dec;112(12):1017-21. doi: 10.1007/s00347-015-0162-z. German. PMID 26602097